CLINICAL TRIAL: NCT05417555
Title: Modulation of Hippocampal Circuitry and Memory Function with Focused Ultrasound in Amnestic MCI
Brief Title: Low Intensity Focused Ultrasound for Mild Cognitive Impairment and Mild Alzheimer's Disease
Acronym: LIFUP-MCIAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Taylor Kuhn, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#21-000995; 1R01AG073480-01 (NIH); IRB#21-000995 (Other: UCLA)
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; Amnestic Mild Cognitive Disorder; Deep Brain Stimulation; Mild Alzheimer's Disease
Keywords: deep brain stimulation (DBS); transcranial focused ultrasound stimulation (tFUS); memory; low-intensity focused ultrasound pulsation (LIFUP); fMRI; mild cognitive impairment; mci; noninvasive brain stimulation (NIBS); ultrasound; Alzheimer's Disease; Mild Alzheimer's
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Subjects are randomly assigned to one of four treatment dosage conditions: 0, 1, 2 or 3 treatments at each MRI-LIFUP session. After 2 weeks, a second dose is administered with the same dosage level for each subject. Memory assessment occurs once at baseline and remotely after each treatment at the onset of the optimal time window (48 hours) for LIFUP-induced change based on prior data. Finally, after 2 weeks, memory is again assessed. Alternate forms are used for the primary outcome measures to avoid practice effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the participants' caregivers will be blinded to arm assignment. Additionally, the person administering memory testing will be blinded to assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- LIFUP Dose Group 1 (Active Comparator): Administration of low intensity focused ultrasound (LIFUP) dose level 1 to the entorhinal cortex.
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation (LIFUP)
- LIFUP Dose Group 2 (Active Comparator): Administration of low intensity focused ultrasound (LIFUP) dose level 2 to the entorhinal cortex.
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation (LIFUP)
- LIFUP Dose Group 3 (Active Comparator): Administration of low intensity focused ultrasound (LIFUP) dose level 3 to the entorhinal cortex.
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation (LIFUP)
- Sham LIFUP (Sham Comparator): No administration of LIFUP. The device will be affixed to the user's head but not turned on.
  Additionally, if at the end of the study, the treatment has been shown to be effective, placebo subjects will be offered a free session using the optimally effective dose, if they consented to being contacted for this purpose.
  Interventions: Device: Low-Intensity Focused Ultrasound Pulsation (LIFUP)

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound Pulsation (LIFUP) — Low intensity focused ultrasound pulsation will be administered to the left entorhinal cortex at 650kHz, ispta.3 720mW/cm, pulse repetition frequency 100Hz, duty cycle 50%, duration 30s with 30s spacing between sonications, 6 sonications per dose (participants receive 0, 1, 2 or 3 doses depending on group assignment)
  Other Names: transcranial focused ultrasound; tFUS; LIFUP; low intensity focused ultrasound

SUMMARY:
The goal of this study is to investigate whether Low Intensity Focused Ultrasound Pulsation (LIFUP) targeting a part of the brain involved in memory will have an affect on brain activity and whether it may improve memory in people with Mild Cognitive Impairment and Mild Alzheimer's Disease.

The main questions the study seeks to answer are:

1. Can LIFUP increase brain activity in the targeted area?
2. Can LIFUP improve memory in people with MCI and mild AD?
3. Can LIFUP improve connectivity of memory networks in the brain?

Participants in this study will complete MRIs and memory testing, and receive Low Intensity Focused Ultrasound to a part of their brain involved in memory (the entorhinal cortex).

DETAILED DESCRIPTION:
This is a proof of concept trial of Low Intensity Focused Ultrasound Pulsation (LIFUP) targeting the entorhinal cortex in patients with amnestic MCI and Mild Alzheimer's Disease. Participation in the study will entail one Zoom intake session, three in-person sessions and three remote Zoom follow-up sessions over the course of about five weeks. The in-person sessions will take about 5 hours for the first and 3 hours for the following two. The Zoom intake session will take 1-2 hours, and the Zoom follow-up sessions will take about 2 hours each. Participants will be asked to complete questionnaires and tests of learning and memory, have their blood drawn, undergo painless ultrasound stimulation to a part of their brain related to memory, and complete MRI scans of their brain. LIFUP will be administered inside of the MRI scanner, so that we can measure changes in brain activity in real-time.

At the start of the study, you will be randomly assigned to one of four different groups that determines the amount of LIFUP stimulation you will receive. You have an equal chance of being assigned to each group. Participants in one of the three active stimulation groups will receive either 1 dose, 2 doses, or 3 doses of LIFUP at their second in-person session, and will receive the same dose again at their third in-person session. Participants in the placebo group will receive no LIFUP stimulation at either MRI/LIFUP session (in-person visits 2 and 3). However, if at the end of our study, the treatment has been shown to be effective, and you were a placebo subject, we will offer you a free session using the most effective dose.

ELIGIBILITY:
Inclusion Criteria

* Amnestic MCI or Mild Alzheimer's diagnosis
* Age 50-90
* English-speaking
* Ability to provide informed consent
* Normal or corrected-to-normal hearing and vision

Exclusion Criteria

GENERAL

* Participation in another clinical trial
* Active use of immunotherapeutic medications for cognition (Aduhelm, Leqembi, Kisunla)
* Moderate to Severe Alzheimer's
* Inability to provide informed consent

MRI-Related:

* Weight exceeding 275 pounds
* Pregnancy, suspicion of pregnancy, or attempting to become pregnant
* Claustrophobia
* Difficulties during previous MRIs
* Top permanent retainer (bottom only is okay), 5 or more non-removable gold-teeth, metal braces, top spacers, and/or palate expanders
* Any of the following implants: Cardiac Pacemaker, Aneurysm clips, Cochlear implants, Defibrillator, Electrodes or wires, Magnetically-activated device, Spinal cord stimulator, Infusion or insulin pumps, Implanted drug infusion device, Deep brain stimulation device
* Non-removable hairpieces, hairpiece extensions, and/or piercings
* Facial tattoos or permanent makeup
* Metal implants that are MR-incompatible, or where participant is unable to provide sufficient information to determine MR compatibility
* Previous injury by metallic foreign body (e.g., bullet, BB, shrapnel) where the object entered the body and participant lacks doctor's confirmation that it was fully removed

Medical:

* Diagnosis of one or more of the following neurological disorders: Parkinson's disease, Lou Gehrig's disease (ALS), Multiple sclerosis, Cerebral Palsy
* Diagnosis of one or more of the following genetic disorders: Cystic Fibrosis, Sickle Cell Disease
* Diagnosis of one or more of the following psychiatric disorders: Bipolar, Psychosis
* Psychiatric illness that has not been controlled for at least two months (if controlled >2 months, with or without medication, they are not exclusionary)
* Severe lung, liver, heart, and/or kidney disease/s (e.g., heart failure, liver failure, and etc...)
* Diagnosis of thyroid disorder or change of thyroid medication dose within the last 3 months
* Cancer treatment/s with chemotherapy and/or radiation to head and neck, or stage 4 (metastatic) cancer
* Autoimmune disorder or viral infection such as HIV, COVID 19, or hepatitis C that has caused current problems with cognition/memory
* History of substance abuse in the past year
* History of stroke (Transient ischemic attack / mini-stroke not exclusionary if symptoms lasted <1 week)
* History of 2 or more seizures or diagnosis of epilepsy, unless the seizures occurred prior to age 5 alongside a fever.
* History of brain tumor, brain aneurysm, brain hemorrhage, or subdural hematoma (transient ischemic attack not exclusionary)
* Head injury that resulted in loss of consciousness lasting >30 minutes, cognitive issues lasting >18 months, and/or brain abnormalities visible in CT or MRI scan
* Uncontrolled high blood pressure or diabetes
* Heart attack within the last year

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Perfusion Arterial Spin Labeling (ASL) fMRI Signal throughout Brain | 40 minutes
  Perfusion ASL fMRI data will be collected before and after sonication. Analyses will assess the statistical relationship between ASL signal throughout the brain pre and post sonication.
Changes in BOLD-related functional connectivity from baseline in fMRI brain scan to 40 minutes. | 40 minutes
  Primary outcomes for proof of mechanism that may be depicted in the fMRI scans may include changes in BOLD-related functional connectivity increases within the DMN including regions functionally connected to the target.
  BOLD data will be collected before, during, and following LIFUP sonication. Analyses will assess any changes in BOLD signal in the brain following sonication.

SECONDARY OUTCOMES:
Change in Brief Visual Memory Test Scores | 48 hours
  Potential LIFUP-related changes in memory will be assessed via neuropsychological assessments including the Brief Visual Memory Tests (BVMT). Scores range from 0 to 12 and reflect recent, long-term learning, with higher scores indicating better learning.
Change in Verbal Learning Test Scores | 48 hours
  Potential LIFUP-related changes in memory will be assessed via the Rey Auditory Verbal Learning Test (RAVLT) neuropsychological assessment. The RAVLT involves providing participants with 15 unrelated words and asking them to recall the word list. There are 5 trials designed to determine short-term memory and then a 20 minute delay to assess long-term memory. The total words correct in both the short- and long-term trials are used as outcome measures.
Post-hoc biomarker analysis of APOE-4 status as a predictor of tFUS efficacy | Baseline (pre-LIFUP)
  Biomarker post hoc analysis will determine the degree to which blood based biomarkers predict the level of effectiveness of tFUS. Samples are collected before LIFUP is administered.
Post-hoc biomarker analysis of plasma AB42/40 ratio as a predictor of tFUS efficacy | Baseline (pre-LIFUP)
  Biomarker post hoc analysis will determine the degree to which blood based biomarkers predict the level of effectiveness of tFUS. Samples are collected before LIFUP is administered.
  An Aβ42/40 ratio <0.160 suggests a higher-than-normal risk of having of AD and is warranted to support a diagnosis of AD (West et al 2021).
Post-hoc biomarker analysis of plasma ptau as a predictor of tFUS efficacy | Baseline (pre-LIFUP)
  Biomarker post hoc analysis will determine the degree to which blood based biomarkers predict the level of effectiveness of tFUS. Samples are collected before LIFUP is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Y Bookheimer, PhD, Principal Investigator — UCLA Psychiatry & Biobehavioral Sciences; Taylor P Kuhn, PhD, Principal Investigator — UCLA Psychiatry & Biobehavioral Sciences
Locations (1):
- UCLA Semel Institute for Neuroscience and Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hescham S, Lim LW, Jahanshahi A, Blokland A, Temel Y. Deep brain stimulation in dementia-related disorders. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2666-75. doi: 10.1016/j.neubiorev.2013.09.002. Epub 2013 Sep 20. PMID 24060532
- [Background] Lin WT, Chen RC, Lu WW, Liu SH, Yang FY. Protective effects of low-intensity pulsed ultrasound on aluminum-induced cerebral damage in Alzheimer's disease rat model. Sci Rep. 2015 Apr 15;5:9671. doi: 10.1038/srep09671. PMID 25873429
- [Background] Burgess A, Dubey S, Yeung S, Hough O, Eterman N, Aubert I, Hynynen K. Alzheimer disease in a mouse model: MR imaging-guided focused ultrasound targeted to the hippocampus opens the blood-brain barrier and improves pathologic abnormalities and behavior. Radiology. 2014 Dec;273(3):736-45. doi: 10.1148/radiol.14140245. Epub 2014 Sep 15. PMID 25222068
- [Background] Bystritsky A, Korb AS, Douglas PK, Cohen MS, Melega WP, Mulgaonkar AP, DeSalles A, Min BK, Yoo SS. A review of low-intensity focused ultrasound pulsation. Brain Stimul. 2011 Jul;4(3):125-36. doi: 10.1016/j.brs.2011.03.007. Epub 2011 Apr 1. PMID 21777872
- See also: Study Website — http://kuhnlab.io/studies/mci